CLINICAL TRIAL: NCT07216495
Title: Pilot Study of an Aerobic Exercise Intervention During Immune Checkpoint Inhibitor Therapy in Early-stage Triple Negative Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-1303; NCI-2025-07495 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Aerobic Exercise; Early Stage Triple Negative Breast Cancer
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute cardiorespiratory exercise program (Experimental): consisting of 4 in-clinic exercise sessions
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Cardiorespiratory training via treadmill walking for 30 minutes; participants will be supervised by a trained exercise physiologist.

SUMMARY:
To learn if participating in a supervised exercise program can help participants with early-stage TNBC who are receiving ICI therapy before undergoing breast surgery.

DETAILED DESCRIPTION:
Primary Objective To evaluate the feasibility of a supervised cardiorespiratory exercise program in participants with clinical stage 2-3 Triple Negative Breast Cancer (TNBC) undergoing neoadjuvant chemotherapy with immune checkpoint inhibitor therapy.

Secondary Objectives To explore the relationship between cardiorespiratory exercise and circulating immune (CD8+ T) cells in the peripheral blood.

ELIGIBILITY:
Inclusion Criteria

1. female and male participants 18 years or older and willing to provide Informed Consent
2. clinical stage 2 or 3 TNBC (estrogen receptor and progesterone receptor ≤ 10% by immunohistochemistry (IHC) and human epidermal growth factor-2 (HER2) negative (IHC 0, IHC1+, or IHC 2+ with negative fluorescence in situ hybridization))
3. Physically able to walk independently without assistive device and able to march in place for 30 seconds without assistive device
4. Eastern Co-Operative Oncology Group (ECOG) Performance Status 0-1
5. Planned receipt of neoadjuvant chemoICI therapy (carboplatin/taxane in combination with pembrolizumab; taxane options are weekly paclitaxel or every 3 week docetaxel8,46)
6. clearance to participate in the study by the patient's medical oncologist
7. normal bone marrow function
8. able to read/complete study forms/assessments and understand instructions in English

Exclusion criteria:

a) Any physical condition which hinders the ability to safely participate in exercise including: uncontrolled or symptomatic cardiac/respiratory disease (e.g. uncontrolled angina, unusual shortness of breath, congestive heart failure, symptomatic peripheral vascular disease), stroke/myocardial infarction in the past year, fragility fracture, recent or planned orthopedic surgery, or any comorbid condition precluding exercise per the treating physician b) receipt of medications known to influence immune function including corticosteroids (>10 mg prednisone equivalent), other immune-suppressive medication, or beta blockers47 c) Any infection or vaccination within the last 4 weeks d) e) Known HIV-positive participants on combination antiretroviral therapy f) concurrent participation in a therapeutic clinical trial or other exercise program g) pregnant h) medically advised to not exercise i) Unable to walk on a motor-driven treadmill for ~30 minutes at study enrollment j) Adults unable to consent k) No external catheters/drains (e.g., nephrostomy tube, foley catheter). A colostomy or Ileostomy is acceptable.

l) Prior or concurrent non-breast malignancy. Those with prior cancers treated with curative intent are eligible. Participants with known (or history) of hepatitis B positive, or hepatitis C positive infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-04-06 (Estimated); Primary Completion 2028-10-30 (Estimated); Study Completion 2030-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Sukumar, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org